CLINICAL TRIAL: NCT03085927
Title: Mechanisms of Active Music Engagement to Improve Health Outcomes of Children With Cancer and Parents
Acronym: PINPOINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Children's Healthcare of Atlanta (Other); Children's Mercy Hospital Kansas City (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Sheri Robb, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01NR015789 (NIH)
Record Dates: First submitted 2017-02-27; First posted 2017-03-21 (Actual); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Cancer
Keywords: music therapy; neoplasms; play; children; parents
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1-Active Music Engagement (Experimental): Three 45-minute sessions with a board-certified music therapist delivered over three days. Sessions are delivered in a private setting during in-patient hospitalization. During the first visit, parent and child will receive information on common responses of young children to cancer treatment and how parents can use music play activities to support their child during treatment. The music therapist will lead parent and child in a variety of music play activities. Parent and child will receive a music kit that includes items such as hand-held rhythm instruments, puppets, and a music CD. During the second and third visit the music therapist will lead parent and child child through the music play activities, answer questions, and make suggestions for using these activities in the hospital and at home.
  Interventions: Behavioral: Active Music Engagement
- Arm II- Audio-Storybooks (Experimental): Three 45-minute sessions with a board-certified music therapist delivered over three days. Sessions are delivered in a private setting during in-patient hospitalization. Each session children/parents will choose and listen to one of three illustrated children's books with audio recorded narration.
  Interventions: Behavioral: Audio Storybooks

INTERVENTIONS:
Behavioral: Active Music Engagement — Three 45-minute sessions with a board-certified music therapist delivered over three days. Sessions are delivered in a private setting during in-patient hospitalization. During the first visit, parent and child will receive information on common responses of young children to cancer treatment and how parents can use music play activities to support their child during treatment. The music therapist will lead parent and child in a variety of music play activities. Parent and child will receive a music kit that includes items such as hand-held rhythm instruments, puppets, and a music CD. During the second and third visit the music therapist will lead parent and child child through the music play activities, answer questions, and make suggestions for using these activities in the hospital and at home.
  Arms: Arm 1-Active Music Engagement
Behavioral: Audio Storybooks — Three 45-minute sessions with a board-certified music therapist delivered over three days. Sessions are delivered in a private setting during in-patient hospitalization. Each session children/parents will choose and listen to one of three illustrated children's books with audio recorded narration.
  Arms: Arm II- Audio-Storybooks

SUMMARY:
Music therapy, a frequently used arts-based therapy, has become standard palliative care in many pediatric and adult hospitals; however, few studies have examined the mechanisms by which music therapy interventions work. This study investigates behavioral, social, and psychological factors that may explain how an Active Music Engagement (AME) intervention (i.e., an interactive, music-based play intervention) works to manage emotional distress and improve positive health outcomes in parents and young children with cancer during treatment. Findings will provide scientific and clinically relevant practice knowledge to guide delivery of music therapy as a complementary therapy.

DETAILED DESCRIPTION:
Music therapy, a frequently used arts-based therapy, has become standard palliative care in many pediatric and adult hospitals; however, few studies have examined mechanisms by which music therapy interventions work.Based on the Contextual Support Model of Music Therapy, the investigators developed and tested the Active Music Engagement (AME) intervention, establishing it as a feasible and acceptable intervention that reduces emotional distress in young children (ages 3-8) hospitalized for cancer treatment.Emotional distress in young children with cancer during acute treatment and their parents is a prevalent,persistent problem associated with physical symptom distress and diminished quality of life and family function. The music therapist-led AME uses music-based play and parent education/support (music play resource kit; tip sheets), is easy to implement, and teaches parents/children how to therapeutically use a familiar activity to manage distress. The purpose of this two group randomized controlled trial is to identify behavioral, sociological, and psychological variables contributing to positive outcomes observed in previous AME studies (i.e., mediators) and identify for whom the intervention works (i.e., moderators). The investigators will examine proximal mediators of child engagement and parent-child interaction and distal mediators of perceived family normalcy, parent confidence (self-efficacy) about their ability to support their child during treatment, and independent parent/child use of music and play activities to manage distress during hospitalization. The investigators hypothesize these factors mediate change in outcomes of child emotional distress, physical symptom distress, and quality of life; parent emotional/traumatic distress and quality of life; and family function. Specific aims are to examine: 1) effects of proximal and distal mediators of AME on young child/parent outcomes; 2) moderators of AME on young child/parent distress; 3) explore child physical symptom distress (pain, fatigue, nausea) in mediation and moderation models. Child/parent dyads (n=184) will be stratified by age and randomized in blocks of 6 to AME or audio-storybooks; each group will receive three 45-minute sessions with a credentialed music therapist for 3 consecutive days with data collection at baseline, post-intervention, and 30 days later. Mediation effects will be estimated using ANCOVA, fitting appropriate mediation models using MPlus and then testing indirect effects using the percentile bootstrap approach to estimate indirect effect. Moderation effects will be tested by including appropriate interaction terms of the potential moderator with the intervention indicator in our models.

ELIGIBILITY:
Inclusion Criteria (Child/Parent):

* Children ages 3-8 years inclusive.
* Expected treatment course for at least 3 days to receive chemotherapy and/or radiation therapy.
* A consistent parent who can be present for all sessions.

Exclusion Criteria (Child/Parent):

* Child and/or parent do not speak English.
* Child has a significant cognitive impairment that hinders participation (based on physician judgment).

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheri L Robb, PhD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robb SL, Clair AA, Watanabe M, Monahan PO, Azzouz F, Stouffer JW, Ebberts A, Darsie E, Whitmer C, Walker J, Nelson K, Hanson-Abromeit D, Lane D, Hannan A. A non-randomized [corrected] controlled trial of the active music engagement (AME) intervention on children with cancer. Psychooncology. 2008 Jul;17(7):699-708. doi: 10.1002/pon.1301. PMID 18033724
- [Background] Robb SL, Haase JE, Perkins SM, Haut PR, Henley AK, Knafl KA, Tong Y. Pilot Randomized Trial of Active Music Engagement Intervention Parent Delivery for Young Children With Cancer. J Pediatr Psychol. 2017 Mar 1;42(2):208-219. doi: 10.1093/jpepsy/jsw050. PMID 27289068
- [Background] Robb SL. The effect of therapeutic music interventions on the behavior of hospitalized children in isolation: developing a contextual support model of music therapy. J Music Ther. 2000 Summer;37(2):118-46. doi: 10.1093/jmt/37.2.118. PMID 10932125
- [Derived] Robb SL, Stegenga K, Perkins SM, Stump TE, Moody KM, Henley AK, MacLean J, Jacob SA, Delgado D, Haut PR. Mediators and Moderators of Active Music Engagement to Reduce Traumatic Stress Symptoms and Improve Well-being in Parents of Young Children With Cancer. Integr Cancer Ther. 2023 Jan-Dec;22:15347354231218266. doi: 10.1177/15347354231218266. PMID 38145309

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited as dyads (child/parent) at 4 sites from September of 2016 through February of 2020. The first participant was enrolled on September 26, 2016 and the last participant was enrolled on February 20, 2020.
Pre-assignment Details: Participants in this study were enrolled as a dyad (child/parent). Totals listed below represent the numbers of dyads enrolled.
  One dyad of the 137 total dyads enrolled came off study prior to completing baseline measures due to the child's toxicity/side effects of cancer treatment.
Period: Overall Study
Arm/Group | Arm 1-Active Music Engagement | Arm II- Audio-Storybooks
Started (Numbers listed reflect child/parents in a dyad. Arm 1=138 individuals Arm 2=134) | 69 | 67
Study Sessions (Arm 1=130 individuals Arm 2=126 individuals) | 65 (Off Study reasons: Child toxicity/side effects (n=1) Dyad withdrew (n=1) Dyad lost to follow-up (n=2)) | 63 (Off Study reasons: Dyad withdrew (n=3) Dyad became ineligible (n=1))
Time 2 Measures (Arm 1=130 individuals Arm 2=124 individuals) | 65 | 62 (Off Study reasons: Dyad withdrew (n=1))
Completed (Arm 1=126 individuals Arm 2=122 individuals) | 63 (Off Study reasons: Death of child (n=1) Dyad lost to follow up (n=1)) | 61 (Off Study reason: Dyad lost to follow up (n=1))
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 3 | 1
Not completed — Death | 1 | 0
Not completed — Child Toxicity/Side Effects of Treatment | 1 | 0
Not completed — Dyad Became Ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Population: Parents and Children were enrolled as dyads and engaged in sessions together. Some of the outcome measures reflect the children, some the parents, and some both members of the dyad.
Groups:
- Arm 1-Active Music Engagement (Children); Arm 1-Active Music Engagement (Parents): Three 45-minute sessions with a board-certified music therapist delivered over three days. Sessions are delivered in a private setting during in-patient hospitalization. During the first visit, parent and child will receive information on common responses of young children to cancer treatment and how parents can use music play activities to support their child during treatment. The music therapist will lead parent and child in a variety of music play activities. Parent and child will receive a music kit that includes items such as hand-held rhythm instruments, puppets, and a music CD. During the second and third visit the music therapist will lead parent and child child through the music play activities, answer questions, and make suggestions for using these activities in the hospital and at home.
- Arm II- Audio-Storybooks (Children); Arm II- Audio-Storybooks (Parents): Three 45-minute sessions with a board-certified music therapist delivered over three days. Sessions are delivered in a private setting during in-patient hospitalization. Each session children/parents will choose and listen to one of three illustrated children's books with audio recorded narration.
- Total: Total of all reporting groups
Arm/Group | Arm 1-Active Music Engagement (Children) | Arm II- Audio-Storybooks (Children) | Arm 1-Active Music Engagement (Parents) | Arm II- Audio-Storybooks (Parents) | Total
Number analyzed (Participants) | 69 | 67 | 69 | 67 | 272
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 69 | 67 | 0 | 0 | 136
  Between 18 and 65 years | 0 | 0 | 68 | 67 | 135
  >=65 years | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 58 | 61 | 179
  Male | 40 | 36 | 11 | 6 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 13 | 6 | 12 | 39
  Not Hispanic or Latino | 58 | 52 | 59 | 52 | 221
  Unknown or Not Reported | 3 | 2 | 4 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 2 | 3
  Asian | 3 | 0 | 4 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 8 | 7 | 29
  White | 46 | 46 | 48 | 52 | 192
  More than one race | 11 | 12 | 7 | 3 | 33
  Unknown or Not Reported | 2 | 1 | 2 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 69 | 67 | 69 | 67 | 272
Family Normalcy [Mean (Standard Deviation); unit: score on a scale] — Family Normalcy is assessed through The Family Management Measure (FaMM) - Family Life Difficulty Subscale includes 14-items rated on a 5-point Likert-type scale. Subscale items address parents' perceptions of the extent to which having a child with a chronic condition makes family life difficult. Higher values indicate more difficulty managing the condition. Score range 14 - 70.
  score on a scale | NA (NA) — Measures completed by parents once for dyads (parent + child). | NA (NA) — Measures completed by parents once for dyads (parent + child). | 36.0 (10.5) | 37.1 (9.7) | 36.6 (10.1)
Parent Self Efficacy [Mean (Standard Deviation); unit: score on a scale] — Parent Self-Efficacy is assessed through the Parental Beliefs Scale (PBS) for Hospitalized Children, a 20-item scale that measures parental beliefs about their confidence in anticipating changes in their hospitalized child's behavior and confidence in their parental role during hospitalization. Scores range from 20-100, with higher scores indicating more positive beliefs.
  score on a scale | NA (NA) — Measures completed by parents for each dyad (parent + child) | NA (NA) — Measures completed by parents for each dyad (parent + child) | 78.3 (10.0) | 80.1 (11.3) | 79.2 (10.7)
Child Emotional Distress [Mean (Standard Deviation); unit: score on a scale] — Child Emotional Distress is assessed through the Child Health Questionnaire (CHQ-PF98) Mental Health Subscale (Landgraf et al., 1999). This subscale consists of 16 items rated on a 5-point Likert-scale. Scores range from 16 to 80 with lower scores indicating better mental health.
  score on a scale | NA (NA) — Measures completed by parents once for each dyad (parent + child) | NA (NA) — Measures completed by parents once for each dyad (parent + child) | 28.6 (14.1) | 28.6 (12.8) | 28.6 (13.4)
Child Quality of Life [Mean (Standard Deviation); unit: score on a scale] — Child Quality of Life is assessed through the KINDL Questionnaire for Measuring Health-Related Quality of Life in Children. The KINDL consists of 24 parent-report items rated on a 5-point Likert-scale for each subscale. Scores range from 20-100 with higher scores indicating better quality of life.
  score on a scale | NA (NA) — Measures completed by parents once for each dyad (parent + child). | NA (NA) — Measures completed by parents once for each dyad (parent + child). | 70.2 (14.7) | 71.1 (13.3) | 70.6 (14.0)
Parent Emotional and Traumatic Distress [Mean (Standard Deviation); unit: score on a scale] — Parent Emotional and Traumatic Distress was assessed through the Profile of Mood States - Short Form (POMS-SF) which measures mood disturbance. There are 37 items which respondents rate on a 5-point Likert scale. Scores range from 0 to 148 with higher scores indicating greater mood disturbance.
  score on a scale | NA (NA) — Measures completed by parents once for dyads (parent + child). | NA (NA) — Measures completed by parents once for dyads (parent + child). | 51.6 (28.3) | 52.8 (29.3) | 52.2 (28.7)
Stress Symptoms [Mean (Standard Deviation); unit: score on a scale] — Stress Symptoms assessed through the Impact of Events Scale-Revised (IES-R), a 22-item measure that measures traumatic stress symptoms in response to a traumatic event that is specified in the instructions. Parents respond to each item using a 5-point Likert scale. Scores range from 0 to 12 with higher scores indicating greater traumatic stress symptoms.
  score on a scale | NA (NA) — Measures completed by parents once for dyads (parent + child). | NA (NA) — Measures completed by parents once for dyads (parent + child). | 3.4 (2.7) | 3.6 (2.5) | 3.5 (2.6)
Parent Quality of Life [Mean (Standard Deviation); unit: score on a scale] — Parent Quality of Life is assessed through the Index of Well-being, a 9-item semantic differential scale describing present life using adjective extremes. Scores range from 7 to 63 with higher scores meaning greater well-being.
  score on a scale | NA (NA) — Measures completed by parents once for each dyad (parent + child). | NA (NA) — Measures completed by parents once for each dyad (parent + child). | 47.2 (11.0) | 48.0 (9.5) | 47.6 (10.2)
Family Function [Mean (Standard Deviation); unit: score on a scale] — Family Function is assessed through the Family Adaptability and Cohesion Scale II (FACES II), a 30-item scale of items rated using a 5-point Likert scale. Scores range from 1 to 5, with higher scores meaning higher family adaptability and cohesion.
  score on a scale | NA (NA) — Measures completed by parents once for each dyad (parent + child). | NA (NA) — Measures completed by parents once for each dyad (parent + child). | 3.9 (0.5) | 3.8 (0.6) | 3.9 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Family Normalcy Perspective - Family Management Measure (FaMM)
Description: Family Normalcy is assessed through The Family Management Measure (FaMM) - Family Life Difficulty Subscale includes 14-items rated on a 5-point Likert-type scale. Subscale items address parents' perceptions of the extent to which having a child with a chronic condition makes family life difficult. Higher values indicate more difficulty managing the condition. Score range 14 - 70.
Time Frame: Time 2(post-session 3 on day 3) and Time 3 (30-days post-session 3, approximately 33 days)
Population: Parent and child participants were enrolled as a dyad. Parents completed all outcome measures for self and for their child as proxy. Arm 1 had 2 parents who did not complete Time 3 measures leaving only 63 participants for analysis. Arm 2 had one parent who did not complete T2 measures leaving 60 participants for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1-Active Music Engagement | Arm II- Audio-Storybooks
Number analyzed (Participants) | 65 | 61
score on a scale
  Time 2: number analyzed (Participants) | 65 | 60
  Time 2 | 35.3 (9.8) | 36.2 (9.5)
  Time 3: number analyzed (Participants) | 63 | 61
  Time 3 | 34.8 (10.1) | 34.3 (8.7)

2. Primary Outcome: Parent Self-Efficacy - Parental Beliefs Scale (PBS).
Description: Parent Self-Efficacy is assessed through the Parental Beliefs Scale (PBS) for Hospitalized Children, a 20-item scale that measures parental beliefs about their confidence in anticipating changes in their hospitalized child's behavior and confidence in their parental role during hospitalization. Scores range from 20-100, with higher scores indicating more positive beliefs.
Time Frame: Time 2(post-session 3 on day 3) and Time 3 (30-days post-session 3, approximately 33 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1-Active Music Engagement | Arm II- Audio-Storybooks
Number analyzed (Participants) | 65 | 61
score on a scale
  Time 2: number analyzed (Participants) | 65 | 60
  Time 2 | 79.0 (9.8) | 81.9 (11.4)
  Time 3: number analyzed (Participants) | 63 | 61
  Time 3 | 81.1 (10.7) | 84.3 (9.7)

3. Primary Outcome: Child Emotional Distress - Child Health Questionnaire (CHQ)
Description: Child Emotional Distress is assessed through the Child Health Questionnaire (CHQ-PF98) Mental Health Subscale (Landgraf et al., 1999). This subscale consists of 16 items rated on a 5-point Likert-scale. Scores range from 16 to 80 with lower scores indicating better mental health.
Time Frame: Time 2(post-session 3 on day 3) and Time 3 (30-days post-session 3, approximately 33 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1-Active Music Engagement | Arm II- Audio-Storybooks
Number analyzed (Participants) | 65 | 61
score on a scale
  Time 2: number analyzed (Participants) | 65 | 60
  Time 2 | 23.3 (12.0) | 24.0 (13.9)
  Time 3: number analyzed (Participants) | 63 | 61
  Time 3 | 24.1 (11.1) | 22.2 (11.1)

4. Primary Outcome: Child Quality of Life - KINDL.
Description: Child Quality of Life is assessed through the KINDL Questionnaire for Measuring Health-Related Quality of Life in Children. The KINDL consists of 24 parent-report items rated on a 5-point Likert-scale for each subscale. Scores range from 20-100 with higher scores indicating better quality of life.
Time Frame: Time 2(post-session 3 on day 3) and Time 3 (30-days post-session 3, approximately 33 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1-Active Music Engagement | Arm II- Audio-Storybooks
Number analyzed (Participants) | 65 | 61
score on a scale
  Time 2: number analyzed (Participants) | 65 | 60
  Time 2 | 67.6 (13.1) | 69.1 (15.7)
  Time 3: number analyzed (Participants) | 63 | 61
  Time 3 | 70.6 (14.7) | 71.7 (15.7)

5. Primary Outcome: Parent Emotional and Traumatic Stress Symptoms - Profile of Mood States-Short Form (POMS).
Description: Parent Emotional and Traumatic Distress was assessed through the Profile of Mood States - Short Form (POMS-SF) which measures mood disturbance. There are 37 items which respondents rate on a 5-point Likert scale. Scores range from 0 to 148 with higher scores indicating greater mood disturbance.
Time Frame: Time 2(post-session 3 on day 3) and Time 3 (30-days post-session 3, approximately 33 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1-Active Music Engagement | Arm II- Audio-Storybooks
Number analyzed (Participants) | 65 | 61
score on a scale
  Time 2: number analyzed (Participants) | 65 | 60
  Time 2 | 38.0 (22.6) | 42.1 (25.6)
  Time 3: number analyzed (Participants) | 62 | 61
  Time 3 | 42.9 (29.2) | 43.4 (28.4)

6. Primary Outcome: Parent Emotional and Traumatic Stress Symptoms - Impact of Events Scale-Revised (IES-R)
Description: Stress Symptoms assessed through the Impact of Events Scale-Revised (IES-R), a 22-item measure that measures traumatic stress symptoms in response to a traumatic event that is specified in the instructions. Parents respond to each item using a 5-point Likert scale. Scores range from 0 to 12 with higher scores indicating greater traumatic stress symptoms.
Time Frame: Time 2(post-session 3 on day 3) and Time 3 (30-days post-session 3, approximately 33 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1-Active Music Engagement | Arm II- Audio-Storybooks
Number analyzed (Participants) | 65 | 61
score on a scale
  Time 2: number analyzed (Participants) | 65 | 60
  Time 2 | 2.5 (2.2) | 2.5 (2.2)
  Time 3: number analyzed (Participants) | 63 | 61
  Time 3 | 4.7 (4.7) | 4.9 (4.6)

7. Primary Outcome: Parent Quality of Life - Index of Well Being.
Description: Parent Quality of Life is assessed through the Index of Well-being, a 9-item semantic differential scale describing present life using adjective extremes. Scores range from 7 to 63 with higher scores meaning greater well-being.
Time Frame: Time 2(post-session 3 on day 3) and Time 3 (30-days post-session 3, approximately 33 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1-Active Music Engagement | Arm II- Audio-Storybooks
Number analyzed (Participants) | 65 | 61
score on a scale
  Time 2: number analyzed (Participants) | 65 | 60
  Time 2 | 47.6 (10.1) | 47.9 (10.3)
  Time 3: number analyzed (Participants) | 62 | 61
  Time 3 | 48.2 (10.9) | 46.9 (11.2)

8. Primary Outcome: Family Function - Family Adaptability and Cohesion Scale (FACES II).
Description: Family Function is assessed through the Family Adaptability and Cohesion Scale II (FACES II), a 30-item scale of items rated using a 5-point Likert scale. Scores range from 1 to 5, with higher scores meaning higher family adaptability and cohesion.
Time Frame: Time 2(post-session 3 on day 3) and Time 3 (30-days post-session 3, approximately 33 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1-Active Music Engagement | Arm II- Audio-Storybooks
Number analyzed (Participants) | 65 | 61
score on a scale
  Time 2: number analyzed (Participants) | 65 | 60
  Time 2 | 35.3 (9.8) | 36.2 (9.5)
  Time 3: number analyzed (Participants) | 63 | 61
  Time 3 | 34.8 (10.1) | 34.3 (8.7)

ADVERSE EVENTS:
Time Frame: 33 days (Time 1 through Time 3)
Description: The child in the child/parent dyad passed away before Time 3 therefore we took the dyad off study and did not collect Time 3 data.
Groups:
- Arm 1 Parent-Active Music Engagement; Arm 1 Child-Active Music Engagement: Three 45-minute sessions with a board-certified music therapist delivered over three days. Sessions are delivered in a private setting during in-patient hospitalization. During the first visit, parent and child will receive information on common responses of young children to cancer treatment and how parents can use music play activities to support their child during treatment. The music therapist will lead parent and child in a variety of music play activities. Parent and child will receive a music kit that includes items such as hand-held rhythm instruments, puppets, and a music CD. During the second and third visit the music therapist will lead parent and child child through the music play activities, answer questions, and make suggestions for using these activities in the hospital and at home.
- Arm II Parent- Audio-Storybooks; Arm II Child-Audio Storybooks: Three 45-minute sessions with a board-certified music therapist delivered over three days. Sessions are delivered in a private setting during in-patient hospitalization. Each session children/parents will choose and listen to one of three illustrated children's books with audio recorded narration.
  Audio Storybooks: Three 45-minute sessions with a board-certified music therapist delivered over three days. Sessions are delivered in a private setting during in-patient hospitalization. Each session children/parents will choose and listen to one of three illustrated children's books with audio recorded narration.
Arm/Group | Arm 1 Parent-Active Music Engagement | Arm II Parent- Audio-Storybooks | Arm 1 Child-Active Music Engagement | Arm II Child-Audio Storybooks
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/67 | 1/69 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/67 | 0/69 | 0/67
Other Adverse Events (participants affected / at risk) | 0/69 | 0/67 | 0/69 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT03085927/Prot_SAP_001.pdf
  • Informed Consent Form (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT03085927/ICF_000.pdf